CLINICAL TRIAL: NCT05251545
Title: Pulmonary Vein Isolation Using High Power - Short Duration Versus Ablation Index: a Prospective Randomized Trial
Brief Title: Randomized Trial: High Power Short Duration Versus Ablation Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Bosch Medical Center (Other)
Responsible Party: Principal Investigator, Peter Ong, MD, Consultant Cardiologist (in German: Oberarzt), Robert Bosch Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: High power - short duration
Record Dates: First submitted 2022-01-04; First posted 2022-02-22 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Atrial Fibrillation Paroxysmal; Catheter Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High power - short duration (Active Comparator): Pulmonary vein isolation with high power settings of 45 Watts
  Interventions: Other: Pulmonary vein isolation
- Standard energy (Active Comparator): Pulmonary vein isolation with standard power settings (30 Watts)
  Interventions: Other: Pulmonary vein isolation

INTERVENTIONS:
Other: Pulmonary vein isolation — Comparison of power levels in catheter ablation in regard of single procedure success rate (freedom of any atrial arrhythmia with a duration of more than 30 sec. 45 Watts versus standard power levels (30 Watts).

SUMMARY:
The single procedure success rates of durable pulmonary vein isolation (PVI) for paroxysmal atrial fibrillation (PAF) varies between 80 and 90 %.

This prospective, randomized study investigated the efficacy of pulmonary vein isolation with RF-energy following the CLOSE protocol with standard energy application (30 Watts) versus PVI with RF-energy with high power settings (45 Watts).

DETAILED DESCRIPTION:
A total number of 176 patients undergoing de-novo catheter ablation for paroxysmal AF are planned to be randomized to two different treatment arms. In group-A patients, PVI was performed with RF-energy with standard power settings of 30 Watts in a temperature-controlled mode.

The ablation procedure in group B was performed with RF-energy with higher power settings of 45 Watts. In both groups the ablation is performed with ablation index (AI) and following the CLOSE protocol (AI and ≤ 6 mm interlesion distance using a surround flow catheter, Biosense Webster Thermocool STSF).

A total of 88 patients are planned to be randomized into each group, the follow-up period will be 12 months after the first procedure.

The primary endpoint is freedom of all atrial arrhythmias after one procedure. The secondary endpoint is procedural time. The third endpoint is safety.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal atrial fibrillation
* written informed consent

Exclusion Criteria:

* inability to obtain written informed consent
* persistent atrial fibrillation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Single procedure success rate, identified by 48-hours Holder-ECGs every three months | 1 year
  Freedom of any atrial arrhythmia of more than 30 sec during a follow-up period of 12 months after the first procedure.

SECONDARY OUTCOMES:
Procedural data | 1 year
  procedural time

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ong, Prof, Principal Investigator — Robert Bosch Medical Campus
Locations (1):
- Robert Bosch Medical Center, Stuttgart, Germany

IPD SHARING:
Plan to Share IPD: No